CLINICAL TRIAL: NCT06083792
Title: ICP Threshold of Severe Traunatic Brain Injury After Decompressive Craniectomy
Brief Title: ICP Threshold After Decompressive Craniectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K202307-17
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe traumatic brain injury (sTBI) is a critical disease of public health importance. Increased intracranial play a significant role in the secondary injury of TBI. Reducing the ICP is helpful in reducing the mortality of sTBI. The threshold of ICP for sTBI has been suggested. The threshold of ICP for sTBI after decompressive craniectomy is not clear.

DETAILED DESCRIPTION:
240 sTBI patients who meet the inclusion criteria will be enrolled in the present study.

All sTBI patients will be screened. If meeting the including criteria, the investigators will contact the family, explain the study, and send a consent form for review.

After obtaining written consent from the family, the ICP and blood pressure will be monitored continuously until retraction of ICP sensor. A mean ICP of each patient will be calculated. The neurological outcome will be assessed at 180 days after injury. A threshold for ICP after decompressive craniectomy will be derived by analyzing the association between mean ICP and neurological outcome.

ELIGIBILITY:
Inclusion Criteria:

* history of traumatic brain injury age: 18-80 years admission GCS score≤8 admitting to hospital with 24 hours after injury received decompressive craniectomy received invasive ICP monitoring

Exclusion Criteria:

* refuse follow-up received operation before admitting to hospital received cardio-pulmonary resuscitation after injury disturbance of consciousness caused by non-traumatic reasons prior history of traumatic brain injury or stroke expected lifetime less than 180 days admitting to other ongoing study systemic disease: uremia, liver cirrhosis, malignant tumor, mental disease, drug or alcohol dependence

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 240 patients
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-10-08 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Modified Glasgow Outcome score | 180 days after injury
  neurological outcome

CONTACTS AND LOCATIONS:
Overall Officials: Yan Qu, Principal Investigator — Tang-Du Hospital

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR